CLINICAL TRIAL: NCT04481919
Title: A Randomized Trial of Protocolized Diuretic Therapy Compared to Standard Care in Emergency Department Patients With Acute Heart Failure
Brief Title: Randomized Controlled Trial of urinE chemiStry Guided aCute heArt faiLure treATmEnt (ESCALATE)
Acronym: ESCALATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sean Collins, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190690
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Acute Heart Failure
Keywords: Diuretic Therapy; Emergency Department
MeSH Terms: conditions — Heart Failure; Emergencies

STUDY DESIGN:
Intervention Model Description: Two-arm comparison of structured usual care vs urinary sodium guided diuresis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blinded study of guideline-based care compared with a protocolized diuretic strategy using urinary sodium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protocolized spot urine sodium guided diuretic therapy (Active Comparator): Patients will have a spot urine sodium and urine creatinine obtained. The urine and creatinine results will be input into the diuretic calculator and the diuretic dose will be chosen based on daily goals for urine output and net negative fluid balance. Performed 3 times per day, diuretic dosing will be individualized based on the proportion of 24-hour diuresis achieved since the prior IV diuretic dose. Every 24 hours new goals for urine output and net negative fluid balance are established based on the study and treatment team's assessment of residual congestion until protocol completion.
  Interventions: Drug: Protocolized diuretic therapy
- Guideline-based care (No Intervention): Patients will be placed on guideline-based diuretic dosing consistent with usual practice. The initial dose will be two times their home dose and will be subsequently adjusted by the treating team based on renal function and symptom severity. The treating team can increase or decrease the frequency and dose of diuretic based on urine output and clinical assessment. Patients in this arm also have urine collected 3 times per day by the bedside nurse to mirror the intervention arm.

INTERVENTIONS:
Drug: Protocolized diuretic therapy — The urine sodium, urine creatinine and serum creatinine results will be input into the diuretic calculator and the diuretic dose will be chosen based on daily goals for urine output and net negative fluid balance.
  Arms: Protocolized spot urine sodium guided diuretic therapy

SUMMARY:
This is a randomized trial of protocolized diuretic therapy guided by urinary sodium compared to structured usual care in ED patients with AHF. Participants will be recruited following an initial standard evaluation in the ED and randomized in a 1:1 fashion to structured usual care or protocolized diuretic therapy guided by urinary sodium.

DETAILED DESCRIPTION:
A standardized protocol driven treatment pathway for hospitalized patients started in the first few hours of ED evaluation and utilizing objective measures of diuretic response is needed. The investigators believe this would maximize diuretic efficiency, facilitate quicker resolution of congestion, avoid WHF and prolonged LOS, and reduce AHF readmissions. Propr data suggests low urine sodium predicts length of stay and outcomes after initial diuretic dosing in the outpatient and inpatient setting. Further, use of our pathway using spot urine sodium to titrate subsequent loop diuretic doses and maximize response in inpatients with AHF has shown compelling improvements in congestion and weight loss. However, a randomized trial is necessary to determine if initiating this protocol ,started in the ED, will improve AHF outcomes relative to structured usual care. Specifically, the investigators hypothesize use of spot urine sodium guided diuretic therapy will result in significant improvement in days of benefit over the 14 days after randomization. Days of benefit combines patient symptoms captured by global clinical status with clinical state quantifying the need for hospitalization and IV diuresis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Emergency Department diagnosis of Acute Heart Failure (AHF)
* Any one of the following:

  i. Chest radiograph or lung ultrasound consistent with AHF ii. Jugular venous distension iii. Pulmonary rales on auscultation iv. Lower extremity edema v. S3 gallop
* > 10 pounds of volume overload physician estimate or historical dry weight
* IV diuretic ordered or planned to be during first 24 hours of ED or inpatient stay

Exclusion Criteria:

* End Stage Renal Disease (ESRD) requiring dialysis
* Need for immediate intubation
* Acute Coronary Syndrome - presentation consistent with myocardial ischemia AND new ST-Segment elevation/depression
* Temperature > 100.5ºF
* End Stage Heart Failure: transplant list or ventricular assist device
* Concurrent use of ototoxic medications including intravenous aminoglycosides and cisplatin
* Systolic Blood Pressure < 90 mmHg at time of consent
* LV outflow obstruction, severe uncorrected stenotic valvular disease or severe restrictive cardiomyopathy
* Greater than 2 doses of IV diuretic administered at the time of screening from the time of the hospital presentation leading to this admission (outside hospital time is included)
* Severe, uncorrected serum electrolyte abnormalities at the time of consent (serum potassium <3.0 mEq/L, magnesium <1.0 mEq/L or sodium <125 or >150 mEq/l)
* Lack of informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Status Score | From the time of randomization through day 14
  Daily composite of the clinical state and global clinical status (GCS), expressed as an integer ranging in value from 0 (deceased) to 15 (outpatient; best possible GCS).

SECONDARY OUTCOMES:
Inpatient clinical congestion | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  Daily orthodema score
Cardiorenal Death and AHF Readmission | within 30 days of hospital discharge
  Cardiorenal death and Acute Heart Failure Readmission
Global clinical status (GCS) | from the time of randomization through 14 days after randomization
  measured daily using a continuous scale of 1-100
Change in natriuretic peptides | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  Blood measurement
Net fluid loss | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  difference between fluid input and urine output in ml
Total urine output | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  cumulative urine output in ml
Weight Loss | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  cumulative weight loss in pounds
Home days | within 30 days from randomization
  Those days not in the hospital, rehab or a skilled nursing facility from the time of randomization through day 30
Subclinical ototoxicity | at two time points: 1) the day of randomization and 2) the next calendar day after protocolized IV diuretics are stopped
  As measured by shoebox audiometry with a significant change in hearing threshold (dB) across frequencies from 250-8000 Hz
Cumulative natriuresis | from the time of randomization through the end of protocolized diuretics, approximately 14 days
  cumulative sodium excretion estimated using the NRPE (based on spot urine creatinine and sodium)
Average daily natriuresis | from the time of randomization through the end of protocolized diuretics, approximately 14 days
  mean daily sodium excretion estimated using the NRPE (based on spot urine creatinine and sodium)

OTHER OUTCOMES:
Dyspnea score | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  measured daily using a continuous scale from 1-100
Change in Kidney injury biomarkers | from the time of randomization through the end of protocolized IV diuretics, approximately 14 days
  changes in the urinary tubular injury markers such as KIM-1 and NGAL
Hospital Length of stay | from the ED presentation to hospital discharge, approximately 7 days
  number of days in the hospital
180-day all cause death | within 180 days of hospital discharge
  all-cause death
Hypotension | from the time of randomization through 7 days off protocolized IV diuretics, or discharge
  Incidence of symptomatic (lightheaded, chest pain) hypotension (SBP < 80 mmHg confirmed on 2 successive measurements at least 30 minutes apart)
Acute Kidney Injury Differences in Epithelial sodium channel (ENaC) levels | from the time of randomization through 7 days off protocolized IV diuretics, or discharge
  AKI (defined as a need for renal replacement therapy or KDIGO stage 2 or greater from a serum creatinine at randomization)
Cardiorenal death or Myocardial Infarction (MI) during hospitalization | from the time of randomization through 7 days off protocolized IV diuretics, or discharge
  Cardiorenal death or MI as adjudicated by a clinical events committee
Ototoxicity or tinnitus | from the time of randomization through 7 days off protocolized IV diuretics, or discharge
  Clinically significant ototoxicity or tinnitus as determined by the study team

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. Collins, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - VA Tennessee Valley Health Service, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The Publication Committee will authorize access to study data. Investigators must submit a proposal requesting approval to access our trial data. Our trial will participate in the NHLBI Central Repository for study data and specimens.
  All data access will follow guidelines described in the NHLBI Limited Access Data Policy.
Supporting Information: CSR
Access Criteria: The Publication Committee will authorize access to study data. Investigators must submit a proposal requesting approval to access our trial data. Our trial will participate in the NHLBI Central Repository for study data and specimens.
  All data access will follow guidelines described in the NHLBI Limited Access Data Policy

REFERENCES:
- [Derived] Cox ZL, Siddiqi HK, Stevenson LW, Bales B, Han JH, Hart K, Imhoff B, Ivey-Miranda JB, Jenkins CA, Lindenfeld J, Shotwell MS, Miller KF, Ooi H, Rao VS, Schlendorf K, Self WH, Siew ED, Storrow A, Walsh R, Wrenn JO, Testani JM, Collins SP. Randomized controlled trial of urinE chemiStry guided aCute heArt faiLure treATmEnt (ESCALATE): Rationale and design. Am Heart J. 2023 Nov;265:121-131. doi: 10.1016/j.ahj.2023.07.014. Epub 2023 Aug 6. PMID 37544492